CLINICAL TRIAL: NCT03525509
Title: Investigation of Pharmacokinetics and Pharmacodynamics of Epidural Methadone in Healthy Volunteers
Brief Title: Epidural Methadone in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: simon.haroutounian (Other)
Responsible Party: Sponsor-Investigator, simon.haroutounian, Assistant Professor of Anesthesiology, Chief of Clinical Research for Washington University Pain Center, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 201802099
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Pain, Acute
Keywords: Methadone; Morphine; Quantitative sensory testing; Epidural
MeSH Terms: conditions — Acute Pain | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, crossover design in healthy volunteers
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: At enrollment, each participant will be assigned a study number, which will match a previously prepared computer-generated list of randomization numbers to determine the interventions. Pharmacy staff who prepares blinded syringes of medications for administration will not be involved in medication administration, outcomes assessment, or statistical analysis. The participants and all other study personnel will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epidural methadone (Experimental): A single 4mg epidural bolus of methadone hydrochloride
  Interventions: Drug: Methadone hydrochloride
- Epidural morphine (Active Comparator): A single 4mg epidural bolus of morphine sulfate
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Methadone hydrochloride — Epidural bolus of 4mg of preservative free methadone hydrochloride (4mL of 1mg/mL solution)
  Other Names: Epidural methadone
  Arms: Epidural methadone
Drug: Morphine Sulfate — Epidural bolus of 4mg of preservative free morphine sulfate (4mL of 1mg/mL solution)
  Other Names: Epidural morphine
  Arms: Epidural morphine

SUMMARY:
Epidurally administered opioid pain medications are important tools for postoperative pain control, but each agent has its own limitations. Methadone's properties suggest that it may provide a long duration of pain control with minimal side effects related to spread to the brain or absorption into the blood stream. In this study, the investigators aim to compare the relative pain relieving effects, markers of side effects, and concentrations in the blood of epidurally administered methadone as compared to another long-acting opioid which is commonly administered epidurally, morphine.

DETAILED DESCRIPTION:
Acute postoperative pain control remains a major challenge in healthcare, with a need to balance analgesic effectiveness, patient safety, and cost. Excellent analgesia is a universal clinical imperative, but our current approaches are often inadequate. Epidural opioids can be useful tools, but each carries its own strengths and limitations. Bolus morphine is long lasting but exhibits rostral spread in the cerebrospinal fluid, which raises risks of adverse effects, particularly late-onset respiratory depression. Lipophilic opioids such as fentanyl and sufentanil exhibit selective segmental analgesia but are of short duration due to systemic absorption. As such, they require continuous epidural administration via an indwelling epidural catheter and a pump (patient-controlled or continuous infusion), which has implications for nursing, pain management services, and hospital cost. Methadone's physico-chemical properties suggest that epidural methadone administration would be ideal in providing long-duration analgesia with fewer of the adverse effects seen with medications like morphine.

The aim of this study is to compare the effects of two medications given epidurally: morphine and methadone. We will do so using a randomized, double-blinded, crossover design study. During each of two study visits, participants will receive a single epidural bolus of either morphine or methadone. We will examine the ability of the medication to blunt pain from heat or pressure using quantitative sensory testing at both the dermatome of injection (leg) and a distant dermatome (face); in doing so, we will demonstrate relative segmental versus supraspinal or systemic opioid activity. Additionally, we will assess signs and symptoms of supraspinal opioid activity, which may predispose to adverse effects, and blood concentrations of each medication. Each of the aforementioned measurements will be conducted at multiple points over a 24 hour period. Following a washout period, patients will return for a second visit, at which time the protocol will be repeated using the other medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. Body mass index between 18.5 and 30
3. Good general health with no remarkable medical conditions;
4. Able and willing to provide informed consent.

Exclusion Criteria:

1. Known history of hepatic, renal, and cardiac disease;
2. Known history of diabetes mellitus;
3. Chronic pain;
4. A skin or spine condition preventing safe epidural catheter placement;
5. Current pregnancy or lactation;
6. Known coagulopathy or ongoing anticoagulant use which contraindicates epidural catheter placement;
7. Known allergic reactions to opioids or local anesthetics;
8. History of current or prior substance use disorder or positive screen using the 4-question Simple Screening Instrument for Substance Abuse (SSI-SA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Selective segmental analgesia for heat pain - methadone | 0 -12 hours after medication administration
  The analgesia provided by methadone at a given dermatome will be quantified as the area under the curve (AUC) of the heat pain tolerance threshold versus time curve. The selective segmental analgesic effect of methadone will be measured as difference of the AUC for L3 and V2.

SECONDARY OUTCOMES:
Selective segmental analgesia for heat pain - morphine | 0 -12 hours after medication administration
  The analgesia provided by morphine at a given dermatome will be quantified as the area under the curve (AUC) of the heat pain tolerance threshold versus time curve. The selective segmental analgesic effect of morphine will be measured as difference of the AUC for L3 and V2.
Selective segmental analgesia for pressure pain - methadone | 0 - 12 hours after medication administration
  The analgesia provided by methadone at a given dermatome will be quantified as the area under the curve (AUC) of the pressure pain threshold versus time curve. The selective segmental analgesic effect of methadone will be measured as difference of the AUC for L3 and V2.
Selective segmental analgesia for pressure pain - morphine | 0 - 12 hours after medication administration
  The analgesia provided by morphine at a given dermatome will be quantified as the area under the curve (AUC) of the pressure pain threshold versus time curve. The selective segmental analgesic effect of morphine will be measured as difference of the AUC for L3 and V2.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University in Saint Louis; Yehuda Ginosar, MBBS, Principal Investigator — Washington University in Saint Louis
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shir Y, Rosen G, Zeldin A, Davidson EM. Methadone is safe for treating hospitalized patients with severe pain. Can J Anaesth. 2001 Dec;48(11):1109-13. doi: 10.1007/BF03020377. PMID 11744587
- [Background] Haroutiunian S, Kagan L, Yifrach-Damari I, Davidson E, Ratz Y, Hoffman A. Enhanced antinociceptive efficacy of epidural compared with i.v. methadone in a rat model of thermal nociception. Br J Anaesth. 2014 Jan;112(1):150-8. doi: 10.1093/bja/aet234. Epub 2013 Jul 10. PMID 23842610
- [Background] Bernards CM, Shen DD, Sterling ES, Adkins JE, Risler L, Phillips B, Ummenhofer W. Epidural, cerebrospinal fluid, and plasma pharmacokinetics of epidural opioids (part 1): differences among opioids. Anesthesiology. 2003 Aug;99(2):455-65. doi: 10.1097/00000542-200308000-00029. PMID 12883420
- [Background] Gedney JA, Liu EH. Side-effects of epidural infusions of opioid bupivacaine mixtures. Anaesthesia. 1998 Dec;53(12):1148-55. doi: 10.1046/j.1365-2044.1998.00636.x. PMID 10193215